CLINICAL TRIAL: NCT01008657
Title: Multipolar Radiofrequency Ablation for the Treatment of Hepatocellular Carcinoma Using Classical Intranodular Technique Versus Extra Nodular Technique So-called "No Touch" Technique: A Prospective Randomized Trial
Brief Title: Multipolar Radiofrequency Ablation for Hepatocellular Carcinoma Using Extra Nodular Versus Intranodular Technique
Acronym: ARMCENVIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071213
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Hepatocellular Carcinomas
Keywords: Radiofrequency-Extranodular-Multipolar ablation; Recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- extranodular "no touch" multipolar RFA (Experimental)
  Interventions: Procedure: Radiofrequency ablation
- intranodular multipolar RFA (Active Comparator)
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Percutaneous multipolar radiofrequency ablation.
  Other Names: radiofrequency extranodular or intanodular ablation

SUMMARY:
The primary purpose of the trial is to demonstrate that at least a 40% drop of recurrence rate can be achieve in hepatocellular carcinoma patients treated with no touch multipolar radiofrequency ablation technique compared to those treated with usual intranodular multipolar technique.

DETAILED DESCRIPTION:
206 patients with hepatocellular carcinoma(s) including up to three nodules measuring up to four cm in diameter, will be randomized in two therapeutic legs: multipolar no touch radiofrequency versus multipolar intra nodular radiofrequency. Patients previously treated for hepatocellular carcinoma will not be enrolled in the study. Diagnostic of hepatocellular carcinoma will be based on American Society of Liver Diseases guide line. Early response to the treatment will be assessed one month after the radiofrequency ablation procedures (up to three in case of incomplete necrosis) with dynamic contrast medium enhanced CT or MRI liver examinations. For the follow up dynamic contrast medium enhanced CT or MRI liver examinations will be performed every three months.

The trial will last for 73 months including 45 months for the recruitment of patients. The main criteria of judgement will be the 2-years recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years old, holder of up to 3 nodules less than 4 cm in diameter
* Diagnosis of hepatocellular carcinoma according to American Society of Liver Study non invasive criteria or based on histological proof
* Non invasive diagnosis of cirrhosis according to French Haute Authority of illness guideline or based on histological proof
* No previous treatment for hepatocellular carcinoma
* Multidisciplinary decision of treatment by radiofrequency ablation

Exclusion Criteria:

* Adult patient under guardianship or trusteeship, homeless
* Patient with potentially short term life-threatening serious co-infection (apart from viral B or C, or VIH co-infection)
* Pregnant or breastfeeding woman
* Patient for whom regular follow-up is impossible whatever the cause
* Contra indication to general anaesthesia
* Technical impossibility to perform the procedure under ultrasound guidance
* Boundary of the tumor located at less than 1 cm distance from colonic wall or main biliary tract (main right or left bill ducts and common bill duct)
* Tumor invisible with ultrasound
* Lack of safe percutaneous course which can be planned
* Tumor in which more than four biopsies pass were previously performed (cumulated during one or several previous biopsies sessions)
* Contra indication to perform CT or MRI with contrast medium (GADOLINITE or iodinate) intravenous injection
* Child-Pugh B or C cirrhosis (apart from the transitory liver failures in the setting of acute hepatitis related to alcohol abuse)
* Total detachment of the anterior face of the liver from internal abdominal wall due to abundant ascites.
* Prothrombin activity < 50 %
* Platelet count <40 .10 3/ml
* Platelet dysfunction or congenital impaired blood coagulating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2010-02-09 (Actual); Primary Completion 2016-10-06 (Actual); Study Completion 2016-10-06 (Actual)

PRIMARY OUTCOMES:
2 years global (local+distant) recurrence rate | 2 years

SECONDARY OUTCOMES:
2 years local recurrence rate | 2 years
2 years distant recurrence rate | 2 years
Primary treatment effectiveness (assessed 1 month after completion of treatment course which can include up to 3 radiofrequency ablation (RFA) procedures performed monthly) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Seror, professor, Principal Investigator — Radiology Department, CHU-Jean Verdier
Locations (1):
- Radiology Department, Bondy, France

REFERENCES:
- [Background] Chen MS, Li JQ, Zheng Y, Guo RP, Liang HH, Zhang YQ, Lin XJ, Lau WY. A prospective randomized trial comparing percutaneous local ablative therapy and partial hepatectomy for small hepatocellular carcinoma. Ann Surg. 2006 Mar;243(3):321-8. doi: 10.1097/01.sla.0000201480.65519.b8. PMID 16495695
- [Background] Kotoh K, Enjoji M, Arimura E, Morizono S, Kohjima M, Sakai H, Nakamuta M. Scattered and rapid intrahepatic recurrences after radio frequency ablation for hepatocellular carcinoma. World J Gastroenterol. 2005 Nov 21;11(43):6828-32. doi: 10.3748/wjg.v11.i43.6828. PMID 16425391
- [Background] Seror O, N'Kontchou G, Tin-Tin-Htar M, Barrucand C, Ganne N, Coderc E, Trinchet JC, Sellier N, Beaugrand M. Radiofrequency ablation with internally cooled versus perfused electrodes for the treatment of small hepatocellular carcinoma in patients with cirrhosis. J Vasc Interv Radiol. 2008 May;19(5):718-24. doi: 10.1016/j.jvir.2008.01.007. Epub 2008 Mar 17. PMID 18440461
- [Background] Harrison LE, Koneru B, Baramipour P, Fisher A, Barone A, Wilson D, Dela Torre A, Cho KC, Contractor D, Korogodsky M. Locoregional recurrences are frequent after radiofrequency ablation for hepatocellular carcinoma. J Am Coll Surg. 2003 Nov;197(5):759-64. doi: 10.1016/S1072-7515(03)00750-6. PMID 14585410
- [Background] Mazzaferro V, Battiston C, Perrone S, Pulvirenti A, Regalia E, Romito R, Sarli D, Schiavo M, Garbagnati F, Marchiano A, Spreafico C, Camerini T, Mariani L, Miceli R, Andreola S. Radiofrequency ablation of small hepatocellular carcinoma in cirrhotic patients awaiting liver transplantation: a prospective study. Ann Surg. 2004 Nov;240(5):900-9. doi: 10.1097/01.sla.0000143301.56154.95. PMID 15492574
- [Background] Kotoh K, Morizono S, Kohjima M, Enjoji M, Sakai H, Nakamuta M. Evaluation of liver parenchymal pressure and portal endothelium damage during radio frequency ablation in an in vivo porcine model. Liver Int. 2005 Dec;25(6):1217-23. doi: 10.1111/j.1478-3231.2005.01167.x. PMID 16343075
- [Background] Kotoh K, Nakamuta M, Morizono S, Kohjima M, Arimura E, Fukushima M, Enjoji M, Sakai H, Nawata H. A multi-step, incremental expansion method for radio frequency ablation: optimization of the procedure to prevent increases in intra-tumor pressure and to reduce the ablation time. Liver Int. 2005 Jun;25(3):542-7. doi: 10.1111/j.1478-3231.2005.01051.x. PMID 15910491
- [Background] Nakamuta M, Kohjima M, Morizono S, Yoshimoto T, Miyagi Y, Sakai H, Enjoji M, Kotoh K. Comparison of tissue pressure and ablation time between the LeVeen and cool-tip needle methods. Comp Hepatol. 2006 Dec 21;5:10. doi: 10.1186/1476-5926-5-10. PMID 17181870
- [Background] Okusaka T, Okada S, Ueno H, Ikeda M, Shimada K, Yamamoto J, Kosuge T, Yamasaki S, Fukushima N, Sakamoto M. Satellite lesions in patients with small hepatocellular carcinoma with reference to clinicopathologic features. Cancer. 2002 Nov 1;95(9):1931-7. doi: 10.1002/cncr.10892. PMID 12404287
- [Background] Pawlik TM, Delman KA, Vauthey JN, Nagorney DM, Ng IO, Ikai I, Yamaoka Y, Belghiti J, Lauwers GY, Poon RT, Abdalla EK. Tumor size predicts vascular invasion and histologic grade: Implications for selection of surgical treatment for hepatocellular carcinoma. Liver Transpl. 2005 Sep;11(9):1086-92. doi: 10.1002/lt.20472. PMID 16123959
- [Background] Shi M, Guo RP, Lin XJ, Zhang YQ, Chen MS, Zhang CQ, Lau WY, Li JQ. Partial hepatectomy with wide versus narrow resection margin for solitary hepatocellular carcinoma: a prospective randomized trial. Ann Surg. 2007 Jan;245(1):36-43. doi: 10.1097/01.sla.0000231758.07868.71. PMID 17197963
- [Background] Seror O, N'Kontchou G, Ibraheem M, Ajavon Y, Barrucand C, Ganne N, Coderc E, Trinchet JC, Beaugrand M, Sellier N. Large (>or=5.0-cm) HCCs: multipolar RF ablation with three internally cooled bipolar electrodes--initial experience in 26 patients. Radiology. 2008 Jul;248(1):288-96. doi: 10.1148/radiol.2481071101. Epub 2008 May 15. PMID 18483229
- [Background] Wong IH, Yeo W, Leung T, Lau WY, Johnson PJ. Circulating tumor cell mRNAs in peripheral blood from hepatocellular carcinoma patients under radiotherapy, surgical resection or chemotherapy: a quantitative evaluation. Cancer Lett. 2001 Jun 26;167(2):183-91. doi: 10.1016/s0304-3835(01)00455-4. PMID 11369140